CLINICAL TRIAL: NCT00887926
Title: An Open-label, Dose Escalation, Phase I Study of IMC-EB10 in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Study of IMC-EB10 in Participant With Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13959; CP17-0801 (Other: ImClone, LLC); I5C-IE-JEBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Myeloid Leukemia
Keywords: AML; Leukemia; Acute Myeloid Leukemia; Antibodies, Monoclonal
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia; Leukemia, Myeloid, Acute | interventions — IMC-EB10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-EB10 5 milligrams/kilogram (mg/kg) (Experimental): All participants will receive intravenous infusions of IMC-EB10, with the dose depending on which cohort they are enrolled into.
  Interventions: Biological: IMC-EB10

INTERVENTIONS:
Biological: IMC-EB10 — Cohort 1 will receive IMC-EB10 intravenously for 3 weekly infusions, followed by a 1-week observation period. The starting dose in Cohort 1 will be 5 mg/kg. After all participants in Cohort 1 complete the first cycle of therapy, dose escalation for subsequent cohorts will proceed as follows: Cohort 2 - 10 mg/kg, Cohort 3 - 20 mg/kg, Cohort 4 - 30 mg/kg. Participants who experience a dose-limiting toxicity (DLT) will not receive further IMC-EB10 treatment, but will continue to be followed on the protocol. Participants may continue to receive IMC-EB10 therapy, in the absence of treatment failure, treatment intolerance, or other withdrawal criteria for additional 28-day cycles at the same dose that they initially received. Dosing for Cycle 2 and beyond will be administered on Days 1, 8, 15, and 22 of a 28-day treatment cycle
  Other Names: LY3012218

SUMMARY:
The purpose of this study is to determine if IMC-EB10 is safe for participants with leukemia, and also to determine the best dose of IMC-EB10 to give to participants.

DETAILED DESCRIPTION:
The purpose of this study is to define the maximum tolerated dose (MTD) and the pharmacokinetic (PK) profile of the anti-FMS-like tyrosine kinase 3 (FLT3) monoclonal antibody IMC-EB10, administered weekly in participant with acute lymphoblastic leukemia (AML) who have failed to achieve complete remission to a standard induction regimen, relapsed after response to previous antileukemia therapy, or are not eligible for potentially curative or approved salvage options.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has acute myeloid leukemia in the bone marrow or blood that has relapsed with or without a prior complete remission
2. The participant is not regarded to be a candidate for a potentially curative, higher priority treatment for acute myeloid leukemia
3. The participant has resolution of all clinically significant toxic effects of any prior antitumor therapy and any other study-specific clinical or laboratory parameter specified in the entry criteria
4. The participant has not had major surgery, an open biopsy, a significant injury, and/or prior antitumor therapy (except antileukemia therapy) within 21 days prior to the first infusion of IMC-EB10
5. The participant has an Eastern Cooperative Oncology Group (ECOG)performance status of 0, 1, or 2 at study entry.
6. The participant is age 18 years or older
7. The participant has a life expectancy of >3 months
8. The participant has adequate liver and kidney function, as defined in the entry criteria
9. The participant is using an effective contraception (per the institutional standard), if procreative potential exists
10. The participant is able to give written informed consent
11. The participant is willing and able to comply with study procedures, scheduled visits, and treatment plans

Exclusion Criteria:

1. The participant has had prior allogenic or autologous stem cell transplant within <3 months of the first infusion of IMC-EB10
2. The participant has had an organ transplant (nonhematologic) within 3 years of study entry
3. The participant has active central nervous system leukemia
4. The participant has extramedullary disease without peripheral/and or bone marrow involvement
5. The participant is disease-free from a previous or concurrent malignancy for a period ≤ 1 year. A participant who has basal cell carcinoma or carcinoma in situ of the cervix will not be excluded from the study
6. The participant is currently receiving antileukemia therapy. Concurrent treatment with hydroxyurea is permitted
7. The participant has uncontrolled intercurrent illness as specified in the study entry criteria
8. The participant is receiving chronic steroid or other immunosuppressive medications. Occasional use of steroid-containing medications for, for example (e.g.), asthma exacerbation or for skin lesions, is permitted
9. The participant is receiving full-dose heparin (including low molecular weight heparin) or warfarin. [The participant is permitted to use low-dose warfarin to maintain patency of preexisting, permanent, indwelling intravenous (I.V.) catheters.]
10. The participant is pregnant (confirmed by urine or serum pregnancy test) or breast feeding
11. The participant has received treatment with monoclonal antibodies within 6 weeks prior to first infusion of IMC-EB10
12. The participant has a history of clinically significant allergic reactions to monoclonal antibodies or other therapeutic proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - ImClone Investigational Site, Columbus, Ohio
  - ImClone Investigational Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant Flow is reporting enrolled participants who discontinued from the study. Participants who died or had progressive disease (PD) were considered to have completed the study.
Groups:
- Cohort 1 - 5mg/kg IMC-EB10 (LY3012218): IMC-EB10: 5 milligrams/kilogram (mg/kg) administered intravenously (IV) on Days 1, 8, and 15 of Cycle 1 (28-day cycle) and Days 1, 8, 15, and 22 of subsequent 28-day cycles.
- Cohort 2 - 10 mg/kg IMC-EB10: IMC-EB10: 10 mg/kg administered IV on Days 1, 8, and 15 of Cycle 1 (28-day cycle) and Days 1, 8, 15, and 22 of subsequent 28-day cycles.
- Cohort 3 - 20 mg/kg IMC-EB10: IMC-EB10: 20 mg/kg administered IV on Days 1, 8, and 15 of Cycle 1 (28-day cycle) and Days 1, 8, 15, and 22 of subsequent 28-day cycles.
- Cohort 4 - 30 mg/kg IMC-EB10: IMC-EB10: 30 mg/kg administered IV on Days 1, 8, and 15 of Cycle 1 (28-day cycle) and Days 1, 8, 15, and 22 of subsequent 28-day cycles.
Period: Overall Study
Arm/Group | Cohort 1 - 5mg/kg IMC-EB10 (LY3012218) | Cohort 2 - 10 mg/kg IMC-EB10 | Cohort 3 - 20 mg/kg IMC-EB10 | Cohort 4 - 30 mg/kg IMC-EB10
Started | 3 | 14 | 3 | 5
Received at Least 1 Dose of Study Drug | 3 | 13 | 3 | 5
Completed | 3 | 13 | 3 | 5
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Cohort 1 - 5mg/kg IMC-EB10: IMC-EB10: 5 mg/kg administered IV on Days 1, 8, and 15 of Cycle 1 (28-day cycle) and Days 1, 8, 15, and 22 of subsequent 28-day cycles.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 5mg/kg IMC-EB10 | Cohort 2 - 10 mg/kg IMC-EB10 | Cohort 3 - 20 mg/kg IMC-EB10 | Cohort 4 - 30 mg/kg IMC-EB10 | Total
Number analyzed (Participants) | 3 | 13 | 3 | 5 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (5.97) | 63.9 (18.52) | 74.8 (4.45) | 60.3 (16.91) | 65.0 (15.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 1 | 1 | 10
  Male | 3 | 5 | 2 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 10 | 3 | 3 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 13 | 3 | 5 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerate Dose (MTD) of IMC-EB10
Description: MTD is defined as the dose preceding the dose level at which 2 participants experienced a dose limiting toxicity (DLT) during Cycle 1. DLT is defined using National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (NCI-CTCAE v 3.0): (1) any Grade 3 or 4 toxicity that is clearly not attributable to leukemia [for example (e.g.) a type of end-organ failure that is infrequently encountered in acute myeloid leukemia (AML)] and is possibly, probably, or definitely attributable to IMC-EB10 in the judgment of the investigator; and (2) any Grade 3 or 4 toxicity that is clearly not attributable to a co-medication (e.g., prolonged neutropenia that is not attributable to hydroxyurea).
Time Frame: Cycle 1 (28-day cycle)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: mg/kg
Groups:
- IMC-EB10 5 to 30 mg/kg: Participants received either 5, 10, 20 or 30 mg/kg of IMC-EB10 IV on Days 1, 8, and 15 of Cycle 1 (28-day cycle).
Arm/Group | IMC-EB10 5 to 30 mg/kg
Number analyzed (Participants) | 24
mg/kg | NA — The MTD was below the level required for efficacy and the study was terminated early. Therefore, due to insufficient number of participants with events, 30 mg/kg was not fully expanded and the recommended MTD could not be calculated

2. Secondary Outcome: Pharmacokinetic (PK): Maximum Concentration (Cmax)
Time Frame: Cycle 1 Week 1: predose, immediately after infusion, and 1.5, 2, 4, 8, 24, 96, and 168 h after infusion ends, and Cycle 1 Week 3: predose, immediately after infusion, and 1.5, 2, 4, 8, 24, 48, 96,168, 240 and 336 h after infusion ends (28-day cycles)
Population: All randomized participants with Cmax results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Arm/Group | Cohort 1 - 5mg/kg IMC-EB10 | Cohort 2 - 10 mg/kg IMC-EB10 | Cohort 3 - 20 mg/kg IMC-EB10 | Cohort 4 - 30 mg/kg IMC-EB10
Number analyzed (Participants) | 3 | 11 | 3 | 4
micrograms/milliliter (µg/mL)
  Week 1 | 129 (25) | 254 (35) | 896 (30) | 927 (38)
  Week 3: number analyzed (Participants) | 3 | 7 | 3 | 3
  Week 3 | 119 (24) | 781 (66) | 1520 (9) | 1770 (74)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Last Measurable Concentration [AUC(0-last)]
Time Frame: Cycle 1 Week 1: predose, immediately after infusion, and at 1.5, 2, 4, 8, 24, 96 and 168 h after infusion ends (28-day cycle)
Population: All randomized participants with AUC(0-last) results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms * hours/milliliter (µg*h/mL)
Arm/Group | Cohort 1 - 5mg/kg IMC-EB10 | Cohort 2 - 10 mg/kg IMC-EB10 | Cohort 3 - 20 mg/kg IMC-EB10 | Cohort 4 - 30 mg/kg IMC-EB10
Number analyzed (Participants) | 3 | 10 | 3 | 3
micrograms * hours/milliliter (µg*h/mL) | 9090 (39) | 23300 (27) | 71800 (40) | 77200 (69)

4. Secondary Outcome: PK: Area Under the Concentration Time Curve During the Dosing Interval (AUCtau) Where Tau is 168 Hours
Time Frame: Cycle 1 Week 3: predose, immediately after infusion and at 1.5, 2, 4, 8, 24, 48, 96,168, 240 and 336 h after infusion ends (28-day cycle)
Population: All randomized participants with AUCtau results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 1 - 5mg/kg IMC-EB10 | Cohort 2 - 10 mg/kg IMC-EB10 | Cohort 3 - 20 mg/kg IMC-EB10 | Cohort 4 - 30 mg/kg IMC-EB10
Number analyzed (Participants) | 2 | 5 | 3 | 2
µg*h/mL | NA (NA) — The Geometric Mean and Geometric Coefficient of Variation was not estimated because of small number of participants with evaluable data (n=2). Individual participant data not provided for data privacy reasons. | 72500 (41) | 108000 (39) | NA (NA) — The Geometric Mean and Geometric Coefficient of Variation was not estimated because of small number of participants with evaluable data (n=2). Individual participant data not provided for data privacy reasons.

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) (Safety Profile of IMC-EB10)
Description: Clinically significant events were defined as serious adverse events (SAEs) and other non-serious AEs regardless of causality. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module
Time Frame: 8 weeks and 30-day post-treatment follow-up
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Cohort 1 5mg/kg IMC-EB10: IMC-EB10: 5 mg/kg administered IV on Days 1, 8, and 15 of Cycle 1 (28-day cycle) and Days 1, 8, 15, and 22 of subsequent 28-day cycles.
Arm/Group | Cohort 1 5mg/kg IMC-EB10 | Cohort 2 - 10 mg/kg IMC-EB10 | Cohort 3 - 20 mg/kg IMC-EB10 | Cohort 4 - 30 mg/kg IMC-EB10
Number analyzed (Participants) | 3 | 13 | 3 | 5
participants
  SAEs | 1 | 7 | 1 | 3
  Other Non-Serious AEs | 3 | 11 | 3 | 5

6. Secondary Outcome: Number of Participants With Anti-IMC-EB10 Antibodies
Description: A participant is considered positive for antibodies against IMC-EB10 if their blood sample exhibited a post-treatment antibody level that exceeds the positive upper cut point determined from the anti-IMC-EB10 level in healthy untreated individuals. A participant was considered to have an anti-IMC-EB10 response if there are 2 consecutive positive samples or if the final sample tested is positive.
Time Frame: Cycle 1, Weeks 1 and 3 and Cycle 2, Week 1: predose (28-day cycles)
Population: Zero participants were analyzed. The study was discontinued early due to lack of efficacy and no data was collected.
Arm/Group | Cohort 1 - 5mg/kg IMC-EB10 | Cohort 2 - 10 mg/kg IMC-EB10 | Cohort 3 - 20 mg/kg IMC-EB10 | Cohort 4 - 30 mg/kg IMC-EB10
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Antileukemic Complete Response (CR) or Partial Response (PR)
Description: Assessment of antileukemic response was based on hematologic response criteria. PR defined as >1000/microliter (µL) neutrophils and ≥100000/µL platelets in peripheral blood; a decrease of ≥50% in the pretreatment percentage of blasts to 5% to 25% in the bone marrow aspirate or a value of ≤5% blasts if Auer rods are present. Cytogenetic CR defined as normal cytogenetic findings. Molecular CR defined as negative findings for minimal residual disease by automated quantitative Reverse-Transcription-Polymerase Chain Reaction (RT-PCR) and multidimensional flow cytometry. Morphologic CR with incomplete blood count recovery defined as ≤5% blasts (containing no Auer rods) in a bone marrow aspirate with spicules; neutrophil count < 1000/µL or platelets <100000/mL in peripheral blood or no extramedullary leukemia present.
Time Frame: 4 weeks
Population: All randomized participants who received at least 1 dose of study drug.No anti-leukemic responses were observed as there were no responders due to high rate of treatment failures and were not evaluable.
Measure: Number; unit: participants
Arm/Group | Cohort 1 - 5mg/kg IMC-EB10 | Cohort 2 - 10 mg/kg IMC-EB10 | Cohort 3 - 20 mg/kg IMC-EB10 | Cohort 4 - 30 mg/kg IMC-EB10
Number analyzed (Participants) | 3 | 13 | 3 | 5
participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Feline McDonough Sarcoma (FMS)-Like Tyrosine Kinase 3 (FLT3) Response
Description: FLT3 response to IMC-EB10 is defined as wild type, internal tandem duplications (ITD) mutations and other mutations.
Time Frame: Week 4 and Week 8
Population: All randomized participants who received at least 1 dose of study drug. No tyrosine kinase responses were observed as there were no responders due to high rate of treatment failures and were not evaluable.
Measure: Number; unit: participants
Arm/Group | Cohort 1 5mg/kg IMC-EB10 | Cohort 2 - 10 mg/kg IMC-EB10 | Cohort 3 - 20 mg/kg IMC-EB10 | Cohort 4 - 30 mg/kg IMC-EB10
Number analyzed (Participants) | 3 | 13 | 3 | 5
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cohort 1 - 5mg/kg IMC-EB10 | Cohort 2 - 10 mg/kg IMC-EB10 | Cohort 3 - 20 mg/kg IMC-EB10 | Cohort 4 - 30 mg/kg IMC-EB10
Serious Adverse Events (participants affected / at risk) | 1/3 | 7/13 | 1/3 | 3/5
Other Adverse Events (participants affected / at risk) | 3/3 | 11/13 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 5mg/kg IMC-EB10 (N=3) | Cohort 2 - 10 mg/kg IMC-EB10 (N=13) | Cohort 3 - 20 mg/kg IMC-EB10 (N=3) | Cohort 4 - 30 mg/kg IMC-EB10 (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 5mg/kg IMC-EB10 (N=3) | Cohort 2 - 10 mg/kg IMC-EB10 (N=13) | Cohort 3 - 20 mg/kg IMC-EB10 (N=3) | Cohort 4 - 30 mg/kg IMC-EB10 (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 6 (7) | 1 (1) | 2 (3)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Conjunctival pallor (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Because development of IMC-EB10 was put on hold due to lack of efficacy analyses were not carried out as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.